CLINICAL TRIAL: NCT07344818
Title: An Open and Dose-escalation Early Clinical Study of CD19 and CD20 CAR-T Cell Therapy for Relapsed or Refractory Aggressive B-cell Lymphoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Hebei Senlang Biotechnology Co., LTD (Unknown)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Associate Chief Physician, Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19+CD20 dual CAR-T
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: R/R Aggressive B-cell Lymphoma
Keywords: CD19+CD20 dual CAR-T; B-NHL; CAR-T
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: A 3+3 dose-escalation design will be conducted across different dose levels (2E6/kg, 4E6/kg, 6E6/kg), followed by an expansion study after determination of the RP2D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells therapy (Experimental): eligible patients will be treated with CD19+CD20 dual CAR-T cells
  Interventions: Biological: CAR-T cell therapy

INTERVENTIONS:
Biological: CAR-T cell therapy — autologous CD19+CD20 dual CAR-T cells, single injection

SUMMARY:
To observe the efficacy and safety of dual-target chimeric antigen receptor T cells in the treatment of refractory or relapsed aggressive B-cell lymphoma

DETAILED DESCRIPTION:
In this study, anti-CD19 and anti-CD20 dual target CAR-T cell therapy will be explored for patients with relapsed/refractory aggressive B-cell lymphoma. In this study, the 3+3 dose climbing mode will be used to explore the safety and efficacy of dual-target CAR-T cells in r/r B-NHL therapy at different doses. The RP2D dose will be determined after the relevant data is summarized。

ELIGIBILITY:
Inclusion Criteria:

1. The subject or his/her legal guardian is able to understand and voluntarily sign the informed consent form (ICF).
2. Male or female subjects aged ≥18 years at the time of signing the ICF.
3. An expected life expectancy of at least 12 weeks.
4. An ECOG performance status of 0-2 at the time of signing the ICF.
5. A diagnosis of relapsed or refractory aggressive B-cell lymphoma at the time of signing the ICF. Subjects must have previously received treatment with anthracycline-containing chemotherapy and rituximab (or other CD20-targeted agents), and must have experienced relapse or progression after at least two prior lines of therapy or autologous hematopoietic stem cell transplantation (ASCT).
6. Presence of measurable positive lesions as defined by the Lugano criteria.
7. Lymphoma lesions confirmed by biopsy to screening demonstrating expression of CD19 and/or CD20.
8. Adequate major organ function.
9. contraception.

Exclusion Criteria:

1. Lymphoma involving only the central nervous system (CNS) (except for secondary CNS lymphoma).
2. History of CNS disorders.
3. History of autoimmune disease requiring systemic immunosuppressive therapy within 4 weeks prior to signing the ICF.
4. Presence of any uncontrolled active infection at the time of signing the ICF or within 2 weeks prior to leukapheresis, requiring antibiotic, antiviral, or antifungal treatment.
5. Evidence of active infection, including: HBV DNA、Positive anti-HCV antibody with detectable HCV RNA、Positive HIV antibody、Positive cytomegalovirus (CMV) DNA、Positive Epstein-Barr virus (EBV) DNA、Positive both treponemal-specific and non-specific serologic tests for syphilis.
6. Clinically significant cardiovascular disease.
7. Known hypersensitivity to any component of the investigational products used in this study.
8. Receipt of any disease-related investigational therapy or other systemic antitumor therapy prior to leukapheresis and within 5 half-lives of the drug.
9. Requirement for systemic corticosteroids (at a dose equivalent to ≥20 mg/day of prednisone) or other immunosuppressive agents within 2 weeks prior to signing the ICF, within 2 weeks prior to leukapheresis, or during the study.
10. Major surgery (excluding routine biopsy) within 4 weeks prior to signing the ICF, or planned major surgery during the study period.
11. History of another primary malignancy within 5 years prior to signing the ICF, except for:

    1. Adequately treated and cured carcinoma in situ of the cervix;
    2. Localized basal cell carcinoma or squamous cell carcinoma of the skin.
12. Receipt of a live attenuated vaccine within 4 weeks prior to signing the ICF, or planned vaccination with a live attenuated vaccine during the screening period.
13. Any condition or complication that, in the investigator's opinion, may affect protocol compliance or make the subject unsuitable for participation in the study.
14. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
the safety of CD19⁺CD20 CAR-T therapy | 1 year after CAR-T cells therapy
  To evaluate the incidence and severity of AEs and SAEs in the treatment of relapsed or refractory CD19 and/or CD20 positive aggressive B-cell lymphoma patients after infused the CD19+CD20 CAR-T cells

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided